CLINICAL TRIAL: NCT05829889
Title: A Comparison of Fractional Flow Reserve- Versus Angiography-Guided Percutaneous Coronary Intervention in Patients With Left Main Coronary Artery Disease
Brief Title: Fractional Flow Reserve Versus Angiography for Treatment-Decision and Evaluation of Significant Left MAIN Coronary Artery Disease
Acronym: FATE-MAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Cardiology, Asan Medical Center Heart Institute, Valvular Heart Disease Center, Ischemic Heart Disease Center, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2023-02
Record Dates: First submitted 2023-03-30; First posted 2023-04-26 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease Left Main; Coronary Artery Disease
Keywords: Fractional Flow Reserve; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FFR-guided Left Main PCI (Experimental)
  Interventions: Procedure: FFR-Guided PCI
- Angiography-Guided PCI (Active Comparator)
  Interventions: Procedure: Angiography-Guided PCI

INTERVENTIONS:
Procedure: FFR-Guided PCI — Fractional Flow Reserve-Guided PCI
  Arms: FFR-guided Left Main PCI
Procedure: Angiography-Guided PCI — Angiography-Guided PCI
  Arms: Angiography-Guided PCI

SUMMARY:
The primary purpose of the study was to determine whether the 2-year probability of major adverse cardiac events (primary composite outcome) differed significantly between patients who underwent angiography-guided Percutaneous Coronary Intervention(PCI) and those who underwent Fractional Flow Reserve(FFR)-guided PCI in patients with Left Main Coronary Artery disease(LMCA).

DETAILED DESCRIPTION:
All participants will be monitored over a span of two years and the time point of the year of last subject last visit. The term "year of last subject last visit" refers to the time point of the last visit for all participants. At this specific time point, event occurrence check will be conducted to determine the occurrence of endpoint events among all participants.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be ≥20 years of age with angina and/or evidence of myocardial ischemia.
2. Significant de novo LMCA disease, defined as ≥ 50% diameter stenosis by visual estimation with or without concomitant non-left main major epicardial coronary artery disease, amenable to PCI with drug-eluting stent(DES) implantation.
3. The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

1. left anterior descending coronary artery (LAD) or left circumflex coronary artery (LCx) chronic total occlusion (CTO)
2. Extremely calcified or tortuous vessels precluding FFR measurement.
3. The presence of complex coronary disease anatomy or lesion characteristics or other cardiac condition(s) which leads the participating interventional cardiologist to believe that PCI is not suitable (i.e. the subject should be managed with coronary artery bypass graft or medical therapy alone).
4. Recent ST Elevation Myocardial Infarction(<7 days prior to randomization).
5. Cardiogenic shock and/or need for mechanical/pharmacologic hemodynamic support.
6. Severe left ventricular dysfunction (ejection fraction <30%).
7. Requirement for other cardiac surgical procedure (e.g., valve replacement or aorta surgery).
8. Contraindication or inability to take aspirin or P2Y12 inhibitors (clopidogrel, ticagrelor, or clopidogrel).
9. Prior PCI of the left main trunk.
10. Prior coronary artery bypass graft surgery.
11. Subjects requiring or who may require additional surgery (cardiac or noncardiac) within 1 year.
12. End-stage renal disease requiring renal replacement therapy.
13. Liver cirrhosis.
14. Pregnant and/or lactating women.
15. Concurrent medical condition with a limited life expectancy of less than 2 years.
16. Subjects who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period. However, where at least one or more conditions are satisfied, it could be an exception according to an investigator's discretion;

1) Participated in the observational study expected no effect on the safety and/or effectiveness evaluation of this trial.

2) Screening failed before any interventional factor is involved.

3) Participated in academic trials like strategic comparison studies conducted under standard therapy provided that there is no additional risk or a specific procedure to a subject and no interference between this trial and other studies.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The composite event rate | 2 years
  Composite event consists of death from any causes, myocardial infarction, or hospitalization for unstable angina, heart failure, or resuscitated cardiac arrest, or repeat revascularization.
  A composite endpoint is an endpoint that is a combination of multiple clinical endpoints. An event is considered to have occurred if any one of several different events is observed.

SECONDARY OUTCOMES:
The event rate of death from any causes | 2 years
The event rate of myocardial infarction | 2 years
  any, spontaneous or procedural myocardial infarction
The event rate of hospitalization for unstable angina, heart failure, or resuscitated cardiac arrest | 2 years
The event rate of repeat revascularization | 2 years
The composite event rate of death or myocardial infarction | 2 years
The event rate of stent thrombosis | 2 years
  Stent thrombosis by Academic Research Consortium (ARC) definition
The event rate of stroke | 2 years
The event rate of bleeding complications | 2 years
  Bleeding Academic Research Consortium [BARC] type 3-5, which indicates severe bleeding
Procedure time | 1 day
Amount of contrast agent used | 1 day
Length of hospital stay | an average of 7 day
The event rate of rehospitalization | 2 years
  Rehospitalization from any, cardiac, or noncardiac causes
Functional class | 7 days(discharge) and 1, 6, 12, 24 months
  Functional class assessed by the Canadian Cardiovascular Society (CCS) Angina Score classification.
  The minimum and maximum values are I and IV respectively and a higher score means a worse outcome.
Change of angina-related quality of life index | 7 days(discharge) and 1, 6, 12, 24 months
  By the Seattle Angina Questionnaire [SAQ].
  the SAQ is a disease-specific patient-reported outcome (PRO) with 5 domains. Lower score represents poor health status and high score represents good health status.
Change of health-related quality of life index | 7 days(discharge) and 1, 6, 12, 24 months
  By the EQ-5D.
  EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol Group. Range 0 - 1 and a higher score of EQ-5D mean low quality of life.
Number of anti-anginal medications | 7 days(discharge) and 1, 6, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Duk-woo Park, MD, Principal Investigator — Asan Medical Center
Locations (48):
- Hong Kong (2):
  - Princess Margret Hospital( HongKong), Hong Kong
  - Queen Mary Hospital, Hong Kong
- Manipal Hospital, Bangalore, India
- Japan (3):
  - Japanese Red Cross Musashino Hospital, Tokyo
  - NTT East Japan Kanto Hospital, Tokyo
  - Tsuchiura Kyodo General Hospital, Tsuchiura
- South Korea (41):
  - Asan Medical Center, Seoul, Songpa-gu
  - Korea University Ansan Hospital, Ansan
  - Hallym University Sacred Heart Hospital, Anyang
  - Bucheon Sejong Hospital, Bucheon-si
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Pusan National University Yangsan Hospital, Busan
  - Changwon Gyeongsang National University Hospital, Changwon
  - Kangwon National University Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Daejeon St. Mary's Hospital, Catholic University of Korea, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - CHA Ilsan Medical Center, Ilsan
  - Ilsan Myongji Hospital, Ilsan
  - Inje University Ilsan Paik Hospital, Ilsan
  - National Health Insurance Service Ilsan Hospital, Ilsan
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Chungnam National University Sejong Hospital, Seongam
  - Seoul National University Bundang Hospital, Seongnam
  - Chung-Ang University Hospital, Seoul
  - Eunpyeong St. Mary's Hospital, Catholic University of Korea, Seoul
  - Hanyang University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Seoul Metropolitan Boramae Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Yeouido St. Mary's Hospital, Catholic University of Korea, Seoul
  - Ajou University Hospital, Suwon
  - St. Vincent's Hospital, Catholic University of Korea, Suwon
  - Ulsan University Hospital, Ulsan
  - Yongin Severance Hospital, Yŏngin
- Cheng Hsin General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided